CLINICAL TRIAL: NCT04693897
Title: To Explore the Effect of beta3-adrenoceptor Agonist on Patients With Overactive Bladder and Develop Its Urinary Biomarker
Brief Title: Effect of beta3-adrenoceptor Agonist on Patients With Overactive Bladder and as a Urinary Biomarker
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ching-Chung Liang, Professor, Chang Gung Memorial Hospital
Other Study IDs: CMRPG3K2051
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Overactive Bladder Syndrome; Detrusor Overactivity
Keywords: Overactive Bladder Syndrome; Mirabegron; Beta3-adrenoceptor agonist; Detrusor Overactivity; Urodynamics; Biomarker
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Overactive bladder with Mirabegron: 100 patients with overactive bladder syndrome, diagnosed according to 2002 ICS diagnosis will undergo 12 weeks of Mirabegron 50mg once daily use. Evaluation include questionnaire survey and urine beta-3 adrenoceptor concentration.
  Interventions: Drug: Mirabegron 50 MG
- Overactive bladder with Solifenacin: 100 patients with overactive bladder syndrome, diagnosed according to 2002 ICS diagnosis will undergo 12 weeks of Solifenacin 5mg once daily use. Evaluation include questionnaire survey and urine beta-3 adrenoceptor concentration.
  Interventions: Drug: Solifenacin Succinate 5 MG
- Urinary tract infection: Urinary samples for beta-3 adrenoceptor concentration of 100 patients with urinary tract infection.
- Control: Urinary samples for beta-3 adrenoceptor concentration of 100 patients without lower urinary tract symptoms.

INTERVENTIONS:
Drug: Mirabegron 50 MG — Mirabegron 50mg once daily given to treatment in patients with overactive bladder syndrome
  Groups: Overactive bladder with Mirabegron
Drug: Solifenacin Succinate 5 MG — Solifenacin 5mg once daily given to treatment in patients with overactive bladder syndrome
  Groups: Overactive bladder with Solifenacin

SUMMARY:
About one to two million women in Taiwan suffers from overactive bladder (OAB). The most commonly used anti-muscarinic drugs have a high rate of side effects. While beta-3 adrenoceptor agonist, Mirabegron, has far fewer side effects, there are no consensus on whether it can be used as first-line treatment. The investigator's preliminary study showed that the concentration of beta-3 adrenoceptor in the urine of OAB patients is higher than that in the normal control group, so comparing urinary beta-3 adrenoceptor concentration of OAB patients before and after treatment may be used as a biomarker of therapeutic effectiveness. The results of this study will be of great help in understanding the effectiveness of Mirabegron and formulating OAB treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis compatible with 2002 ICS for overactive bladder syndrome
* Symptoms persisted for more than 3 months
* Completed pre-treatment urodynamic study
* Has plans for treatment with Mirabegron or Solifenacin due to clinical symptoms
* Patient is willing to cooperate with study including follow up and complete questionnaire surveys

Exclusion Criteria:

* Has stress urinary incontinence
* Pelvic organ prolapse
* Interstitial cystitis
* Constipation
* Gastroesophageal reflux disease
* Prior failed medical treatment for overactive bladder syndrome
* Uncontrolled hypertension
* Glaucoma
* Currently pregnant
* Using other medications for overactive bladder syndrome

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with overactive bladder syndrome for 3 or more months with or without concurrent detrusor overactivity treated as outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in participant's urinary beta-3 adrenoreceptor from baseline to 12 weeks after treatment | 12 weeks
  Concentrations of urinary beta-3 adrenoceptor levels will be analyzed for 1)before and after treatment of patients with overactive bladder syndrome treated with Mirabegron; 2)before and after treatment patients with overactive bladder syndrome treated with Solifenacin; 3)patients with urinary tract infection, and 4)control (subjects without lower urinary tract symptoms).

SECONDARY OUTCOMES:
Effect of treatment with Mirabegron in patients with overactive bladder with or without detrusor overactivity after 12 weeks of treatment | 12 weeks
  Individual participant's change score on Overactive Bladder Symptom Score (OABSS) will be compared between participants treated with Mirabegron with and without detrusor overactivity after 12 weeks of treatment. The OABSS is a validated symptom questionnaire that sums the score of four symptoms (daytime frequency, nighttime frequency, urgency, and urgency incontinence). The total score ranges from 0 to 15, with higher the number, the greater the symptoms are.
Effect of treatment with Mirabegron in patients with overactive bladder with or without detrusor overactivity 6 months after treatment. | 6 months
  Individual participant's change score on Overactive Bladder Symptom Score (OABSS) will be compared between participants treated with Mirabegron with and without detrusor overactivity 6 months after treatment. The OABSS is a validated symptom questionnaire that sums the score of four symptoms (daytime frequency, nighttime frequency, urgency, and urgency incontinence). The total score ranges from 0 to 15, with higher the number, the greater the symptoms are.
Change in impact on the participant's life after treatment with Mirabegron with overactive bladder with or without detrusor overactivity after 12 weeks of treatment. | 12 weeks
  Individual participant's change score on the Overactive Bladder Questionnaire short-form (OAB-q SF) will be compared between participants treated with Mirabegron with and without detrusor overactivity after 12 weeks of treatment. The OAB-q SF assess the impact of OAB symptoms on the patient's life, and consists of symptom-bother and health-related quality of life. The subscales are summed and transformed into scores ranging from 0 to 100; a high symptom-bother score indicates greater symptom severity and a high health-related quality of life scale score indicates higher quality of life.
Change in impact on the participant's life after treatment with Mirabegron with overactive bladder with or without detrusor overactivity 6 months after treatment | 6 months
  Individual participant change score on the Overactive Bladder Questionnaire short-form (OAB-q SF) will be compared between participants treated with Mirabegron with and without detrusor overactivity 6 months after treatment. The OAB-q SF assess the impact of OAB symptoms on the patient's life, and consists of symptom-bother and health-related quality of life. The subscales are summed and transformed into scores ranging from 0 to 100; a high symptom-bother score indicates greater symptom severity and a high health-related quality of life scale score indicates higher quality of life.
Effect on the participant's life after treatment with Mirabegron with overactive bladder with or without detrusor overactivity after 12 weeks of treatment. | 12 weeks
  Individual participant's change score on Short Form Health Survey (SF-12) will be compared between participants treated with Mirabegron with and without detrusor overactivity after 12 weeks of treatment. SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The score is converted to a range of 0 to 100, with high the score indicating a better quality of life.
Effect on the participant's life after treatment with Mirabegron with overactive bladder with or without detrusor overactivity 6 months after treatment. | 6 months
  Individual participant's change score on Short Form Health Survey (SF-12) will be compared between participants treated with Mirabegron with and without detrusor overactivity 6 months after treatment. SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The score is converted to a range of 0 to 100, with high the score indicating a better quality of life.
The participant's subjective measurement of treatment outcome with Mirabegron with overactive bladder with or without detrusor overactivity after 12 weeks of treatment. | 12 weeks
  Individual participant's change score on Global Response Assessment Scale (GRAS) will be compared between participants treated with Mirabegron with and without detrusor overactivity after 12 weeks of treatment. GRAS is a subjective outcome measurement to asses the participant's perception of treatment success. The score is scaled from 0 to 100%, with greater the percentage, the greater improvement of symptoms after treatment is perceived.
The participant's subjective measurement of treatment outcome with Mirabegron with overactive bladder with or without detrusor overactivity 6 months after treatment. | 6 months
  Individual participant's change score on Global Response Assessment Scale (GRAS) will be compared between participants treated with Mirabegron with and without detrusor overactivity 6 months after treatment. GRAS is a subjective outcome measurement to asses the participant's perception of treatment success. The score is scaled from 0 to 100%, with greater the percentage, the greater improvement of symptoms after treatment is perceived.
Comparison of the effect of treatment with Mirabegron and Solifenacin in patients with overactive bladder after 12 weeks of treatment | 12 weeks
  Individual participant's change score on Overactive Bladder Symptom Score (OABSS) will be compared between participants treated with Mirabegron and Solifenacin in patients with overactive bladder after 12 weeks of treatment. The OABSS is a validated symptom questionnaire that sums the score of four symptoms (daytime frequency, nighttime frequency, urgency, and urgency incontinence). The total score ranges from 0 to 15, with higher the number, the greater the symptoms are.
Comparison of the effect of treatment with Mirabegron and Solifenacin in patients with overactive bladder 6 months after treatment. | 6 months
  Individual participant's change score on Overactive Bladder Symptom Score (OABSS) will be compared between participants treated with Mirabegron and Solifenacin in patients with overactive bladder 6 months after treatment. The OABSS is a validated symptom questionnaire that sums the score of four symptoms (daytime frequency, nighttime frequency, urgency, and urgency incontinence). The total score ranges from 0 to 15, with higher the number, the greater the symptoms are.
Comparison of the impact of symptoms on life with Mirabegron and Solifenacin in patients with overactive bladder after 12 weeks of treatment | 12 weeks
  Individual participant change score on the Overactive Bladder Questionnaire short-form (OAB-q SF) will be compared between participants treated with Mirabegron and Solifenacin in patients with overactive bladder after 12 weeks of treatment. The OAB-q SF assess the impact of OAB symptoms on the patient's life, and consists of symptom-bother and health-related quality of life. The subscales are summed and transformed into scores ranging from 0 to 100; a high symptom-bother score indicates greater symptom severity and a high health-related quality of life scale score indicates higher quality of life.
Comparison of the impact of symptoms on life with Mirabegron and Solifenacin in patients with overactive bladder 6 months after treatment | 6 months
  Individual participant change score on the Overactive Bladder Questionnaire short-form (OAB-q SF) will be compared between participants treated with Mirabegron and Solifenacin in patients with overactive bladder 6 months after treatment. The OAB-q SF assess the impact of OAB symptoms on the patient's life, and consists of symptom-bother and health-related quality of life. The subscales are summed and transformed into scores ranging from 0 to 100; a high symptom-bother score indicates greater symptom severity and a high health-related quality of life scale score indicates higher quality of life.
Effect on the participant's life after treatment with Mirabegron and Solifenacin after 12 weeks of treatment. | 12 weeks
  Individual participant's change score on Short Form Health Survey (SF-12) will be compared between participants treated with Mirabegron and Solifenacin after 12 weeks of treatment. SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The score is converted to a range of 0 to 100, with high the score indicating a better quality of life.
Effect on the participant's life after treatment with Mirabegron and Solifenacin 6 months after treatment. | 6 months
  Individual participant's change score on Short Form Health Survey (SF-12) will be compared between participants treated with Mirabegron and Solifenacin 6 months after treatment. SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. The score is converted to a range of 0 to 100, with high the score indicating a better quality of life.
The participant's subjective measurement of treatment outcome with Mirabegron and Solifenacin after 12 weeks of treatment. | 12 weeks
  Individual participant's change score on Global Response Assessment Scale (GRAS) will be compared between participants treated with Mirabegron and Solifenacin after 12 weeks of treatment. GRAS is a subjective outcome measurement to asses the participant's perception of treatment success. The score is scaled from 0 to 100%, with greater the percentage, the greater improvement of symptoms after treatment is perceived.
The participant's subjective measurement of treatment outcome with Mirabegron and Solifenacin 6 months after treatment. | 6 months
  Individual participant's change score on Global Response Assessment Scale (GRAS) will be compared between participants treated with Mirabegron and Solifenacin 6 months after treatment. GRAS is a subjective outcome measurement to asses the participant's perception of treatment success. The score is scaled from 0 to 100%, with greater the percentage, the greater improvement of symptoms after treatment is perceived.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coyne KS, Sexton CC, Kopp ZS, Ebel-Bitoun C, Milsom I, Chapple C. The impact of overactive bladder on mental health, work productivity and health-related quality of life in the UK and Sweden: results from EpiLUTS. BJU Int. 2011 Nov;108(9):1459-71. doi: 10.1111/j.1464-410X.2010.10013.x. Epub 2011 Mar 3. PMID 21371240
- [Result] Jafarabadi M, Jafarabadi L, Shariat M, Rabie Salehi G, Haghollahi F, Rashidi BH. Considering the prominent complaint as a guide in medical therapy for overactive bladder syndrome in women over 45 years. J Obstet Gynaecol Res. 2015 Jan;41(1):120-6. doi: 10.1111/jog.12483. Epub 2014 Nov 5. PMID 25369726
- [Result] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Result] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Result] Chen GD, Lin TL, Hu SW, Chen YC, Lin LY. Prevalence and correlation of urinary incontinence and overactive bladder in Taiwanese women. Neurourol Urodyn. 2003;22(2):109-17. doi: 10.1002/nau.10010. PMID 12579627
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Result] Hung MJ, Ho ES, Shen PS, Sun MJ, Lin AT, Chen GD; Taiwan OAB Club. Urgency is the core symptom of female overactive bladder syndrome, as demonstrated by a statistical analysis. J Urol. 2006 Aug;176(2):636-40. doi: 10.1016/j.juro.2006.03.062. PMID 16813910
- [Result] Andersson KE. Antimuscarinics for treatment of overactive bladder. Lancet Neurol. 2004 Jan;3(1):46-53. doi: 10.1016/s1474-4422(03)00622-7. PMID 14693111
- [Result] Ouslander JG. Management of overactive bladder. N Engl J Med. 2004 Feb 19;350(8):786-99. doi: 10.1056/NEJMra032662. No abstract available. PMID 14973214
- [Result] Luo D, Liu L, Han P, Wei Q, Shen H. Solifenacin for overactive bladder: a systematic review and meta-analysis. Int Urogynecol J. 2012 Aug;23(8):983-91. doi: 10.1007/s00192-011-1641-7. Epub 2012 Feb 7. PMID 22310924
- [Result] Nazir J, Kelleher C, Aballea S, Maman K, Hakimi Z, Mankowski C, Odeyemi I. Comparative efficacy and tolerability of solifenacin 5 mg/day versus other oral antimuscarinic agents in overactive bladder: A systematic literature review and network meta-analysis. Neurourol Urodyn. 2018 Mar;37(3):986-996. doi: 10.1002/nau.23413. Epub 2017 Nov 15. PMID 29140559
- [Result] Cardozo L, Thorpe A, Warner J, Sidhu M. The cost-effectiveness of solifenacin vs fesoterodine, oxybutynin immediate-release, propiverine, tolterodine extended-release and tolterodine immediate-release in the treatment of patients with overactive bladder in the UK National Health Service. BJU Int. 2010 Aug;106(4):506-14. doi: 10.1111/j.1464-410X.2009.09160.x. Epub 2010 Feb 3. PMID 20132203
- [Result] Madhuvrata P, Cody JD, Ellis G, Herbison GP, Hay-Smith EJ. Which anticholinergic drug for overactive bladder symptoms in adults. Cochrane Database Syst Rev. 2012 Jan 18;1:CD005429. doi: 10.1002/14651858.CD005429.pub2. PMID 22258963
- [Result] Chapple CR, Fianu-Jonsson A, Indig M, Khullar V, Rosa J, Scarpa RM, Mistry A, Wright DM, Bolodeoku J; STAR study group. Treatment outcomes in the STAR study: a subanalysis of solifenacin 5 mg and tolterodine ER 4 mg. Eur Urol. 2007 Oct;52(4):1195-203. doi: 10.1016/j.eururo.2007.05.027. Epub 2007 Jun 6. PMID 17574730
- [Result] Speakman M, Khullar V, Mundy A, Odeyemi I, Bolodeoku J. A cost-utility analysis of once daily solifenacin compared to tolterodine in the treatment of overactive bladder syndrome. Curr Med Res Opin. 2008 Aug;24(8):2173-9. doi: 10.1185/03007990802234829. Epub 2008 Jun 18. PMID 18565239
- [Result] Takeda M, Obara K, Mizusawa T, Tomita Y, Arai K, Tsutsui T, Hatano A, Takahashi K, Nomura S. Evidence for beta3-adrenoceptor subtypes in relaxation of the human urinary bladder detrusor: analysis by molecular biological and pharmacological methods. J Pharmacol Exp Ther. 1999 Mar;288(3):1367-73. PMID 10027879
- [Result] Igawa Y, Yamazaki Y, Takeda H, Hayakawa K, Akahane M, Ajisawa Y, Yoneyama T, Nishizawa O, Andersson KE. Functional and molecular biological evidence for a possible beta3-adrenoceptor in the human detrusor muscle. Br J Pharmacol. 1999 Feb;126(3):819-25. doi: 10.1038/sj.bjp.0702358. PMID 10188996
- [Result] Tyagi P, Thomas CA, Yoshimura N, Chancellor MB. Investigations into the presence of functional Beta1, Beta2 and Beta3-adrenoceptors in urothelium and detrusor of human bladder. Int Braz J Urol. 2009 Jan-Feb;35(1):76-83. doi: 10.1590/s1677-55382009000100012. PMID 19254402
- [Result] Otsuka A, Shinbo H, Matsumoto R, Kurita Y, Ozono S. Expression and functional role of beta-adrenoceptors in the human urinary bladder urothelium. Naunyn Schmiedebergs Arch Pharmacol. 2008 Jun;377(4-6):473-81. doi: 10.1007/s00210-008-0274-y. Epub 2008 Mar 1. PMID 18311486
- [Result] Yamaguchi O. Beta3-adrenoceptors in human detrusor muscle. Urology. 2002 May;59(5 Suppl 1):25-9. doi: 10.1016/s0090-4295(01)01635-1. PMID 12007519
- [Result] Aizawa N, Igawa Y, Nishizawa O, Wyndaele JJ. Effects of CL316,243, a beta 3-adrenoceptor agonist, and intravesical prostaglandin E2 on the primary bladder afferent activity of the rat. Neurourol Urodyn. 2010 Jun;29(5):771-6. doi: 10.1002/nau.20826. PMID 19816919
- [Result] Aizawa N, Homma Y, Igawa Y. Effects of mirabegron, a novel beta3-adrenoceptor agonist, on primary bladder afferent activity and bladder microcontractions in rats compared with the effects of oxybutynin. Eur Urol. 2012 Dec;62(6):1165-73. doi: 10.1016/j.eururo.2012.08.056. Epub 2012 Sep 5. PMID 22981677
- [Result] Chen HL, Chen TC, Chang HM, Juan YS, Huang WH, Pan HF, Chang YC, Wu CM, Wang YL, Lee HY. Mirabegron is alternative to antimuscarinic agents for overactive bladder without higher risk in hypertension: a systematic review and meta-analysis. World J Urol. 2018 Aug;36(8):1285-1297. doi: 10.1007/s00345-018-2268-9. Epub 2018 Mar 19. PMID 29556972
- [Result] Vecchioli Scaldazza C, Morosetti C. Comparison of Therapeutic Efficacy and Urodynamic Findings of Solifenacin Succinate versus Mirabegron in Women with Overactive Bladder Syndrome: Results of a Randomized Controlled Study. Urol Int. 2016;97(3):325-329. doi: 10.1159/000445808. Epub 2016 Apr 20. PMID 27092789
- [Result] Kuo HC, Lee KS, Na Y, Sood R, Nakaji S, Kubota Y, Kuroishi K. Results of a randomized, double-blind, parallel-group, placebo- and active-controlled, multicenter study of mirabegron, a beta3-adrenoceptor agonist, in patients with overactive bladder in Asia. Neurourol Urodyn. 2015 Sep;34(7):685-92. doi: 10.1002/nau.22645. Epub 2014 Aug 17. PMID 25130281
- [Result] Hsiao SM, Chang TC, Wu WY, Chen CH, Yu HJ, Lin HH. Comparisons of urodynamic effects, therapeutic efficacy and safety of solifenacin versus tolterodine for female overactive bladder syndrome. J Obstet Gynaecol Res. 2011 Aug;37(8):1084-91. doi: 10.1111/j.1447-0756.2010.01493.x. Epub 2011 Apr 19. PMID 21501328
- [Result] Sheng W, Zhang H, Ruth KH. Could urinary nerve growth factor be a biomarker for overactive bladder? A meta-analysis. Neurourol Urodyn. 2017 Sep;36(7):1703-1710. doi: 10.1002/nau.23210. Epub 2017 Jan 19. PMID 28102552
- [Result] Steers WD, Kolbeck S, Creedon D, Tuttle JB. Nerve growth factor in the urinary bladder of the adult regulates neuronal form and function. J Clin Invest. 1991 Nov;88(5):1709-15. doi: 10.1172/JCI115488. PMID 1939656
- [Result] Clemow DB, Steers WD, Tuttle JB. Stretch-activated signaling of nerve growth factor secretion in bladder and vascular smooth muscle cells from hypertensive and hyperactive rats. J Cell Physiol. 2000 Jun;183(3):289-300. doi: 10.1002/(SICI)1097-4652(200006)183:33.0.CO;2-6. PMID 10797303
- [Result] Liu HT, Kuo HC. Urinary nerve growth factor level could be a potential biomarker for diagnosis of overactive bladder. J Urol. 2008 Jun;179(6):2270-4. doi: 10.1016/j.juro.2008.01.146. Epub 2008 Apr 18. PMID 18423678
- [Result] Liu HT, Kuo HC. Urinary nerve growth factor levels are elevated in patients with overactive bladder and do not significantly increase with bladder distention. Neurourol Urodyn. 2009;28(1):78-81. doi: 10.1002/nau.20599. PMID 19089891
- [Result] Mukerji G, Yiangou Y, Grogono J, Underwood J, Agarwal SK, Khullar V, Anand P. Localization of M2 and M3 muscarinic receptors in human bladder disorders and their clinical correlations. J Urol. 2006 Jul;176(1):367-73. doi: 10.1016/S0022-5347(06)00563-5. PMID 16753445
- [Result] Chuang YC, Fraser MO, Yu Y, Chancellor MB, de Groat WC, Yoshimura N. The role of bladder afferent pathways in bladder hyperactivity induced by the intravesical administration of nerve growth factor. J Urol. 2001 Mar;165(3):975-9. PMID 11176525
- [Result] Liu HT, Chancellor MB, Kuo HC. Decrease of urinary nerve growth factor levels after antimuscarinic therapy in patients with overactive bladder. BJU Int. 2009 Jun;103(12):1668-72. doi: 10.1111/j.1464-410X.2009.08380.x. Epub 2009 Feb 11. PMID 19220267
- [Result] Ciftci S, Ozkurkcugil C, Yilmaz H, Ustuner M, Yavuz U, Yuksekkaya M, Cekmen MB. Urinary nerve growth factor and a variable solifenacin dosage in patients with an overactive bladder. Int Urogynecol J. 2016 Feb;27(2):275-80. doi: 10.1007/s00192-015-2825-3. Epub 2015 Aug 27. PMID 26310546
- [Result] Hashim H, Abrams P. Is the bladder a reliable witness for predicting detrusor overactivity? J Urol. 2006 Jan;175(1):191-4; discussion 194-5. doi: 10.1016/S0022-5347(05)00067-4. PMID 16406907
- [Result] Digesu GA, Khullar V, Cardozo L, Salvatore S. Overactive bladder symptoms: do we need urodynamics? Neurourol Urodyn. 2003;22(2):105-8. doi: 10.1002/nau.10099. PMID 12579626
- [Result] Sekido N, Hinotsu S, Kawai K, Shimazui T, Akaza H. How many uncomplicated male and female overactive bladder patients reveal detrusor overactivity during urodynamic study? Int J Urol. 2006 Oct;13(10):1276-9. doi: 10.1111/j.1442-2042.2006.01558.x. PMID 17010004
- [Result] Giarenis I, Mastoroudes H, Srikrishna S, Robinson D, Cardozo L. Is there a difference between women with or without detrusor overactivity complaining of symptoms of overactive bladder? BJU Int. 2013 Aug;112(4):501-7. doi: 10.1111/j.1464-410X.2012.11652.x. Epub 2013 Mar 4. PMID 23452071
- [Result] Diamond P, Hassonah S, Alarab M, Lovatsis D, Drutz HP. The prevalence of detrusor overactivity amongst patients with symptoms of overactive bladder: a retrospective cohort study. Int Urogynecol J. 2012 Nov;23(11):1577-80. doi: 10.1007/s00192-012-1781-4. Epub 2012 Apr 25. PMID 22531957
- [Result] Jeong SJ, Lee SC, Jeong CW, Hong SK, Byun SS, Lee SE. Clinical and urodynamic differences among women with overactive bladder according to the presence of detrusor overactivity. Int Urogynecol J. 2013 Feb;24(2):255-61. doi: 10.1007/s00192-012-1817-9. Epub 2012 May 16. PMID 22588142
- [Result] Malone-Lee JG, Al-Buheissi S. Does urodynamic verification of overactive bladder determine treatment success? Results from a randomized placebo-controlled study. BJU Int. 2009 Apr;103(7):931-7. doi: 10.1111/j.1464-410X.2009.08361.x. Epub 2009 Mar 5. PMID 19281469
- [Result] Nitti VW, Rovner ES, Bavendam T. Response to fesoterodine in patients with an overactive bladder and urgency urinary incontinence is independent of the urodynamic finding of detrusor overactivity. BJU Int. 2010 May;105(9):1268-75. doi: 10.1111/j.1464-410X.2009.09037.x. Epub 2009 Nov 4. PMID 19889062